CLINICAL TRIAL: NCT01345669
Title: A Randomised, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of Afatinib (BIBW 2992) as Adjuvant Therapy After Chemo-radiotherapy in Primary Unresected Patients With Stage III, IVa, or IVb Loco-regionally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: LUX-Head&Neck 2: A Phase III Trial of Afatinib (BIBW 2992) Versus Placebo for the Treatment of Head and Neck Squamous Cell Cancer After Treatment With Chemo-radiotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1200.131; 2011-000392-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Afatinib

ARMS (2):
- Afatinib (BIBW 2992) (Experimental): Once daily
  Interventions: Drug: Afatinib
- Placebo (Placebo Comparator): Once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Once daily
  Arms: Placebo
Drug: Afatinib — Once daily
  Arms: Afatinib (BIBW 2992)

SUMMARY:
This randomised, double-blind phase III trial will be performed in patients with head and neck squamous cell carcinoma (HNSCC). The objectives of the trial are to compare the efficacy and safety of afatinib (BIBW 2992) with placebo as adjuvant therapy to patients who have received definitive chemo-radiotherapy.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically confirmed loco-regionally advanced head and neck squamous cell carcinoma (HNSCC), stage III to IVb
2. Unresected tumour prior to chemo-radiotherapy (CRT)
3. Concomitant CRT completed prior to randomisation
4. After concomitant platinum-based CRT, no evidence of disease (NED) on clinical and radiographic examinations
5. Eastern cooperative oncology group (ECOG) performance status 0 or 1

Exclusion criteria:

1. Prior treatment with epidermal growth factor receptor (EGFR)-targeted small molecules, EGFR-targeted antibodies, and/or any investigational agents for HNSCC
2. Patients with smoking history of less than or equal to 10 pack years and with primary tumour site of base of tongue and/or tonsil
3. Any other malignancy (except for simultaneous HNSCC primaries, appropriately treated superficial basal cell skin cancer and surgically cured cervical cancer in situ) unless free of disease for at least five years
4. Known pre-existing Interstitial Lung Disease (ILD)
5. Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2011-10-17 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (162):
- United States (15):
  - 1200.131.00171 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1200.131.00181 Boehringer Ingelheim Investigational Site, Orange, California
  - 1200.131.00177 Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - 1200.131.00185 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 1200.131.00173 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1200.131.00176 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1200.131.00182 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1200.131.00175 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 1200.131.00179 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 1200.131.00188 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1200.131.10200 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1200.131.00172 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1200.131.00184 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1200.131.00198 Boehringer Ingelheim Investigational Site, Spokane Valley, Washington
  - 1200.131.00183 Boehringer Ingelheim Investigational Site, Wenatchee, Washington
- Argentina (5):
  - 1200.131.05451 Boehringer Ingelheim Investigational Site, Ciudad Autonoma de Bs As
  - 1200.131.05457 Boehringer Ingelheim Investigational Site, Córdoba
  - 1200.131.05458 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
  - 1200.131.05452 Boehringer Ingelheim Investigational Site, Santa Fe
  - 1200.131.05453 Boehringer Ingelheim Investigational Site, Villa Domínico
- 1200.131.06151 Boehringer Ingelheim Investigational Site, Wooloongabba, Queensland, Australia
- Austria (5):
  - 1200.131.04353 Boehringer Ingelheim Investigational Site, Leoben
  - 1200.131.04357 Boehringer Ingelheim Investigational Site, Linz
  - 1200.131.04355 Boehringer Ingelheim Investigational Site, Salzburg
  - 1200.131.04351 Boehringer Ingelheim Investigational Site, Vienna
  - 1200.131.04359 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (7):
  - 1200.131.03259 Boehringer Ingelheim Investigational Site, Brussels
  - 1200.131.03256 Boehringer Ingelheim Investigational Site, Charleroi
  - 1200.131.03255 Boehringer Ingelheim Investigational Site, Hasselt
  - 1200.131.03253 Boehringer Ingelheim Investigational Site, Kortrijk
  - 1200.131.03252 Boehringer Ingelheim Investigational Site, Liège
  - 1200.131.03254 Boehringer Ingelheim Investigational Site, Liège
  - 1200.131.03258 Boehringer Ingelheim Investigational Site, Namur
- Brazil (6):
  - 1200.131.05554 Boehringer Ingelheim Investigational Site, Barretos
  - 1200.131.05555 Boehringer Ingelheim Investigational Site, Jaú
  - 1200.131.05557 Boehringer Ingelheim Investigational Site, Passo Fundo
  - 1200.131.05553 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1200.131.05551 Boehringer Ingelheim Investigational Site, São Paulo
  - 1200.131.05556 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (6):
  - 1200.131.00152 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1200.131.00157 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1200.131.00151 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 1200.131.00153 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1200.131.00154 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1200.131.00155 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Chile (2):
  - 1200.131.05652 Boehringer Ingelheim Investigational Site, Vina de Mar
  - 1200.131.05651 Boehringer Ingelheim Investigational Site, Viña del Mar
- Czechia (3):
  - 1200.131.04254 Boehringer Ingelheim Investigational Site, Brno
  - 1200.131.04251 Boehringer Ingelheim Investigational Site, Prague
  - 1200.131.04253 Boehringer Ingelheim Investigational Site, Prague
- 1200.131.04551 Boehringer Ingelheim Investigational Site, København Ø, Denmark
- 1200.131.2052 Boehringer Ingelheim Investigational Site, Alexandria, Egypt
- 1200.131.35851 Boehringer Ingelheim Investigational Site, Turku, Finland
- France (12):
  - 1200.131.03353 Boehringer Ingelheim Investigational Site, Le Havre
  - 1200.131.03362 Boehringer Ingelheim Investigational Site, Marseille
  - 1200.131.03359 Boehringer Ingelheim Investigational Site, Nice
  - 1200.131.03365 Boehringer Ingelheim Investigational Site, Orléans
  - 1200.131.03355 Boehringer Ingelheim Investigational Site, Pierre-Bénite
  - 1200.131.03367 Boehringer Ingelheim Investigational Site, Rouen
  - 1200.131.03370 Boehringer Ingelheim Investigational Site, Saint-Cloud
  - 1200.131.03354 Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1200.131.03369 Boehringer Ingelheim Investigational Site, Saint-Priest-en-Jarez
  - 1200.131.03366 Boehringer Ingelheim Investigational Site, Salouël
  - 1200.131.03356 Boehringer Ingelheim Investigational Site, Tours
  - 1200.131.03357 Boehringer Ingelheim Investigational Site, Villejuif
- Germany (10):
  - 1200.131.04954 Boehringer Ingelheim Investigational Site, Essen
  - 1200.131.04961 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1200.131.04953 Boehringer Ingelheim Investigational Site, Hanover
  - 1200.131.04956 Boehringer Ingelheim Investigational Site, Jena
  - 1200.131.04959 Boehringer Ingelheim Investigational Site, Kaiserslautern
  - 1200.131.04951 Boehringer Ingelheim Investigational Site, Leipzig
  - 1200.131.04957 Boehringer Ingelheim Investigational Site, Rostock
  - 1200.131.04964 Boehringer Ingelheim Investigational Site, Trier
  - 1200.131.04963 Boehringer Ingelheim Investigational Site, Ulm
  - 1200.131.04962 Boehringer Ingelheim Investigational Site, Villingen-Schwenningen
- Greece (2):
  - 1200.131.03054 Boehringer Ingelheim Investigational Site, Chaïdári
  - 1200.131.03052 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hungary (5):
  - 1200.131.03651 Boehringer Ingelheim Investigational Site, Budapest
  - 1200.131.03652 Boehringer Ingelheim Investigational Site, Budapest
  - 1200.131.03656 Boehringer Ingelheim Investigational Site, Budpest
  - 1200.131.03654 Boehringer Ingelheim Investigational Site, Debrecen
  - 1200.131.03655 Boehringer Ingelheim Investigational Site, Kecskemét
- India (15):
  - 1200.131.09178 Boehringer Ingelheim Investigational Site, Ahmadābād
  - 1200.131.09165 Boehringer Ingelheim Investigational Site, Bangalore
  - 1200.131.09152 Boehringer Ingelheim Investigational Site, Bikaner
  - 1200.131.09163 Boehringer Ingelheim Investigational Site, Chennai
  - 1200.131.09173 Boehringer Ingelheim Investigational Site, Chennai
  - 1200.131.09179 Boehringer Ingelheim Investigational Site, Delhi
  - 1200.131.09170 Boehringer Ingelheim Investigational Site, Gūrgaon
  - 1200.131.09180 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1200.131.09172 Boehringer Ingelheim Investigational Site, Jaipur
  - 1200.131.09176 Boehringer Ingelheim Investigational Site, Karamsad,Anand, Gujarat
  - 1200.131.09162 Boehringer Ingelheim Investigational Site, Madurai, Tamil Nadu
  - 1200.131.09175 Boehringer Ingelheim Investigational Site, Mazagaon, Mumbai
  - 1200.131.09151 Boehringer Ingelheim Investigational Site, New Delhi
  - 1200.131.09164 Boehringer Ingelheim Investigational Site, Pune
  - 1200.131.09159 Boehringer Ingelheim Investigational Site, Visakhapatnam
- Israel (2):
  - 1200.131.97251 Boehringer Ingelheim Investigational Site, Haifa
  - 1200.131.97253 Boehringer Ingelheim Investigational Site, Petah Tikva
- Italy (4):
  - 1200.131.03957 Boehringer Ingelheim Investigational Site, Confreria (CN)
  - 1200.131.03951 Boehringer Ingelheim Investigational Site, Milan
  - 1200.131.03955 Boehringer Ingelheim Investigational Site, Milan
  - 1200.131.03960 Boehringer Ingelheim Investigational Site, Milan
- Japan (12):
  - 1200.131.08156 Boehringer Ingelheim Investigational Site, Aichi, Nagoya
  - 1200.131.08153 Boehringer Ingelheim Investigational Site, Chiba, Kashiwa
  - 1200.131.08151 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1200.131.08161 Boehringer Ingelheim Investigational Site, Hyogo, Akashi
  - 1200.131.08157 Boehringer Ingelheim Investigational Site, Hyogo, Kobe
  - 1200.131.08159 Boehringer Ingelheim Investigational Site, Kanagawa, Isehara
  - 1200.131.08164 Boehringer Ingelheim Investigational Site, Miyagi, Natori
  - 1200.131.08160 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1200.131.08155 Boehringer Ingelheim Investigational Site, Shizuoka, Sunto-gun
  - 1200.131.08152 Boehringer Ingelheim Investigational Site, Tochigi, Shimotsuke
  - 1200.131.08163 Boehringer Ingelheim Investigational Site, Tokyo, Koto-ku
  - 1200.131.08154 Boehringer Ingelheim Investigational Site, Tokyo, Meguro-ku
- 1200.131.05252 Boehringer Ingelheim Investigational Site, México, Mexico
- Netherlands (3):
  - 1200.131.03152 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1200.131.03153 Boehringer Ingelheim Investigational Site, Leiden
  - 1200.131.03151 Boehringer Ingelheim Investigational Site, Rotterdam
- Portugal (5):
  - 1200.131.35155 Boehringer Ingelheim Investigational Site, Almada
  - 1200.131.35154 Boehringer Ingelheim Investigational Site, Coimbra
  - 1200.131.35152 Boehringer Ingelheim Investigational Site, Evora
  - 1200.131.35153 Boehringer Ingelheim Investigational Site, Lisbon
  - 1200.131.35151 Boehringer Ingelheim Investigational Site, Porto
- Russia (7):
  - 1200.131.00759 Boehringer Ingelheim Investigational Site, Moscow
  - 1200.131.00753 Boehringer Ingelheim Investigational Site, Omsk
  - 1200.131.00760 Boehringer Ingelheim Investigational Site, Pyatigorsk
  - 1200.131.00761 Boehringer Ingelheim Investigational Site, Pyatigorsk
  - 1200.131.00763 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1200.131.00755 Boehringer Ingelheim Investigational Site, Ufa
  - 1200.131.00762 Boehringer Ingelheim Investigational Site, Ufa
- Spain (15):
  - 1200.131.03461 Boehringer Ingelheim Investigational Site, Ávila
  - 1200.131.03451 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.131.03454 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.131.03463 Boehringer Ingelheim Investigational Site, Girona
  - 1200.131.03452 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1200.131.03459 Boehringer Ingelheim Investigational Site, Lugo
  - 1200.131.03457 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.131.03464 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.131.03465 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.131.03456 Boehringer Ingelheim Investigational Site, Málaga
  - 1200.131.03462 Boehringer Ingelheim Investigational Site, Málaga
  - 1200.131.03455 Boehringer Ingelheim Investigational Site, Pamplona
  - 1200.131.03460 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón, Madrid
  - 1200.131.03466 Boehringer Ingelheim Investigational Site, Seville
  - 1200.131.03458 Boehringer Ingelheim Investigational Site, Zaragoza
- Sweden (2):
  - 1200.131.04652 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1200.131.04651 Boehringer Ingelheim Investigational Site, Stockholm
- Switzerland (2):
  - 1200.131.04151 Boehringer Ingelheim Investigational Site, Basel
  - 1200.131.04152 Boehringer Ingelheim Investigational Site, Bern
- Ukraine (2):
  - 1200.131.03854 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1200.131.03851 Boehringer Ingelheim Investigational Site, Kiev
- United Kingdom (10):
  - 1200.131.04456 Boehringer Ingelheim Investigational Site, Denbighshire
  - 1200.131.04455 Boehringer Ingelheim Investigational Site, Edinburgh
  - 1200.131.04459 Boehringer Ingelheim Investigational Site, Exeter
  - 1200.131.04460 Boehringer Ingelheim Investigational Site, Glasgow
  - 1200.131.04453 Boehringer Ingelheim Investigational Site, Leicester
  - 1200.131.04451 Boehringer Ingelheim Investigational Site, London
  - 1200.131.04452 Boehringer Ingelheim Investigational Site, Manchester
  - 1200.131.04454 Boehringer Ingelheim Investigational Site, Sheffield
  - 1200.131.04458 Boehringer Ingelheim Investigational Site, Sutton
  - 1200.131.04457 Boehringer Ingelheim Investigational Site, Whitchurch, Cardiff

REFERENCES:
- [Derived] Burtness B, Haddad R, Dinis J, Trigo J, Yokota T, de Souza Viana L, Romanov I, Vermorken J, Bourhis J, Tahara M, Martins Segalla JG, Psyrri A, Vasilevskaya I, Nangia CS, Chaves-Conde M, Kiyota N, Homma A, Holeckova P, Del Campo JM, Asarawala N, Nicolau UR, Rauch D, Even C, Wang B, Gibson N, Ehrnrooth E, Harrington K, Cohen EEW; LUX-Head & Neck 2 investigators. Afatinib vs Placebo as Adjuvant Therapy After Chemoradiotherapy in Squamous Cell Carcinoma of the Head and Neck: A Randomized Clinical Trial. JAMA Oncol. 2019 Aug 1;5(8):1170-1180. doi: 10.1001/jamaoncol.2019.1146. PMID 31194247
- [Derived] Burtness B, Bourhis JP, Vermorken JB, Harrington KJ, Cohen EE. Afatinib versus placebo as adjuvant therapy after chemoradiation in a double-blind, phase III study (LUX-Head & Neck 2) in patients with primary unresected, clinically intermediate-to-high-risk head and neck cancer: study protocol for a randomized controlled trial. Trials. 2014 Nov 29;15:469. doi: 10.1186/1745-6215-15-469. PMID 25432788

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, placebo-controlled, double-blind, parallel arms, multinational phase III trial in which patients were randomised 2:1 to Afatinib or Placebo.
Groups:
- Afatinib (BIBW 2992): Patient received Afatinib film-coated tablets with starting dose 40 mg (milligram)/day and escalation to 50 mg/day and/or reduction to 40, 30 or 20 mg/day according to absence or presence of drug-related adverse events (AEs), orally, once daily for up to 80 weeks or until recurrence / occurrence of second primary tumour, unacceptable side effects, or other reason necessitating withdrawal.
- Placebo: Patient received placebo matching Afatinib film-coated tablets with matching Afatinib dosage regimen, orally, once daily for up to 80 weeks or until recurrence / occurrence of second primary tumour, unacceptable side effects, or other reason necessitating withdrawal.
Period: Overall Study
Arm/Group | Afatinib (BIBW 2992) | Placebo
Started | 411 | 206
Completed | 124 | 87
Not Completed | 287 | 119
Not completed — Primary tumour recurrence | 53 | 32
Not completed — Second primary tumour | 4 | 3
Not completed — Adverse Event | 63 | 9
Not completed — Protocol Violation | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 52 | 13
Not completed — Other Reasons | 111 | 60

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): Included all patients who were randomised, regardless of taking investigational treatment (as randomised)
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib (BIBW 2992) | Placebo | Total
Number analyzed (Participants) | 411 | 206 | 617
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (8.23) | 57.3 (8.64) | 58.0 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 28 | 89
  Male | 350 | 178 | 528

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: Disease Free Survival defined as the time from randomisation until documented tumour recurrence/ second primary tumour (SPT) or death from any cause, whichever occurred first.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Afatinib (BIBW 2992) | Placebo
Number analyzed (Participants) | 411 | 206
Months | 43.40 [16.82 to NA] — Non calculable because the 75th percentile hasn't been reached | NA [16.69 to NA] — Non calculable because the median hasn't been reached
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Placebo; DFS was analysed using a stratified log-rank test with nodal status (N0- N2a vs. N2b-N3) and Eastern Cooperative Oncology Group (ECOG) performance status (0 vs. 1) being the stratification factors; Test type: Superiority or Other; p = 0.4806, Log Rank; Hazard Ratio (HR) = 1.126, 95% CI 2-sided [0.809 to 1.569] — Hazard ratio (Afatinib vs. Placebo) from Cox proportional hazards model stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3)

2. Secondary Outcome: Disease Free Survival (DFS) Rate at 2 Years
Description: Disease Free Survival (DFS) rate at 2 years. Probability of being disease free at 2 years in percentage is provided based on Kaplan-Meier method.
Time Frame: Up to 2 years
Population: Randomised Set, the number of patients from the randomized set those are disease free (or DFS) at 2 years.
Measure: Number (95% Confidence Interval); unit: Probability (%)
Arm/Group | Afatinib (BIBW 2992) | Placebo
Number analyzed (Participants) | 117 | 76
Probability (%) | 67.2 [61.2 to 72.5] | 73.5 [66.0 to 79.5]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Placebo; Kaplan-Meier (KM) curves were calculated for each treatment group, separately, and the estimates of DFS probabilities from the curves and 95% Confidence interval (CI) (using the Greenwood standard error estimate) were tabulated; Test type: Superiority or Other; p = 0.1610, Log Rank; Difference in Kaplan-Meier estimates = -6.27, 95% CI 2-sided [-15.04 to 2.50] — Difference in Kaplan-Meier estimates of Afatinib vs. Placebo is provided

3. Secondary Outcome: Percentage of Patient Deaths (Overall Survival (OS))
Description: Overall survival (OS), defined as the time from randomisation until death (regardless of cause). Due to the small event rate in both treatment arms caused by the early termination of the trial, the hazard estimate is not interpretable. Hence presented the total randomized and the percentage of patients died.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | Afatinib (BIBW 2992) | Placebo
Number analyzed (Participants) | 411 | 206
Percentage of patients | 15.1 [16.82 to NA] | 11.2 [16.69 to NA]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Placebo; Hazard ratio from Cox proportional hazards model stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Test type: Superiority or Other; p = 0.1301, Log Rank — p-value (two-sided) from log-rank test stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Hazard Ratio (HR) = 1.444, 95% CI 2-sided [0.895 to 2.332]

4. Secondary Outcome: Patients With Improved Health Related Quality of Life (HRQOL)
Description: HRQoL questionnaires focused on 3 scales: Pain scale from H&N35, Swallowing scale from H&N35 and Global health status/QoL scale from C30. Improvement was defined as a score that improved from baseline by at least 10 points (on the 0-100 point scale) at any time during the study. If a patient had not improved, worsening was defined as a 10-point worsening at any time during the study. Patients who had neither improved nor worsened were considered as stable. Percentages of patients with improvement in HRQoL are presented.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Patients
Arm/Group | Afatinib (BIBW 2992) | Placebo
Number analyzed (Participants) | 411 | 206
Percentage of Patients
  Swallowing (Q5-Q8 from QLQ-HN35) | 34.8 [16.82 to NA] | 27.2 [16.69 to NA]
  Pain HN35 (Q1-Q4 from QLQ-HN35) | 33.8 | 26.2
  Global health status/QoL(Q29-Q30 from QLQ-C30) | 33.6 | 38.3
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Placebo; Odds ratio and p-value from logistic regression analysis of 'improved vs. not improved' stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3) for Swallowing (Q5-Q8 from QLQ-HN35); Test type: Superiority or Other; p = 0.0561, Regression, Logistic; Odds Ratio (OR) = 1.431, 95% CI 2-sided [0.991 to 2.068]
Statistical Analysis 2: Comparison: Afatinib (BIBW 2992) vs Placebo; Odds ratio and p-value from logistic regression analysis of 'improved vs. not improved' stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3) for Pain HN35 (Q1-Q4 from QLQ-HN35); Test type: Superiority or Other; p = 0.0523, Regression, Logistic; Odds Ratio (OR) = 1.446, 95% CI 2-sided [0.996 to 2.098]
Statistical Analysis 3: Comparison: Afatinib (BIBW 2992) vs Placebo; Odds ratio and p-value from logistic regression analysis of 'improved vs. not improved' stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3) for Global health status/QoL(Q29-Q30 from QLQ-C30); Test type: Superiority or Other; p = 0.2570, Regression, Logistic; Odds Ratio (OR) = 0.818, 95% CI 2-sided [0.577 to 1.158]

5. Secondary Outcome: Time to Deterioration in Health Related Quality of Life (HRQOL)
Description: HRQoL questionnaires focused on 3 scales: Pain scale from H&N35, Swallowing scale from H&N35 and Global health status/QoL scale from C30. Time to deterioration was defined as the time from randomisation to the first 10-point worsening on the 0-100 point scale. Patients with no deterioration (including those with disease recurrence/SPT) were censored at the last available HRQoL assessment date. Patients with no post-baseline assessments were censored on the day of randomisation.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Afatinib (BIBW 2992) | Placebo
Number analyzed (Participants) | 411 | 206
Months
  Swallowing | 18.43 [3.68 to NA] — Non calculable because the 75th percentile hasn't been reached | 31.44 [3.78 to NA] — Non calculable because the 75th percentile hasn't been reached
  Pain HN35 | 12.06 [1.91 to NA] — Non calculable because the 75th percentile hasn't been reached | 31.08 [3.78 to NA] — Non calculable because the 75th percentile hasn't been reached
  Global health status/QoL | 7.59 [1.87 to NA] — Non calculable because the 75th percentile hasn't been reached | 25.79 [6.21 to NA] — Non calculable because the 75th percentile hasn't been reached
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Placebo; For swallowing scale; Hazard ratio from Cox proportional hazard model stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Test type: Superiority or Other; p = 0.0591, Log Rank — P-value from log-rank test stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Hazard Ratio (HR) = 1.295, 95% CI 2-sided [0.986 to 1.700]
Statistical Analysis 2: Comparison: Afatinib (BIBW 2992) vs Placebo; For pain HN35 scale; Hazard ratio from Cox proportional hazard model stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Test type: Superiority or Other; p = 0.0049, Log Rank — P-value from log-rank test stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Hazard Ratio (HR) = 1.456, 95% CI 2-sided [1.113 to 1.905]
Statistical Analysis 3: Comparison: Afatinib (BIBW 2992) vs Placebo; For global health status/QoL scale; Hazard ratio from Cox proportional hazard model stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Test type: Superiority or Other; p = 0.0002, Log Rank — P-value from log-rank test stratified by baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3); Hazard Ratio (HR) = 1.604, 95% CI 2-sided [1.238 to 2.079]

6. Secondary Outcome: Health Related Quality of Life (HRQOL) Scores Over Time
Description: HRQoL questionnaires focused on 3 scales: Pain scale from H&N35, Swallowing scale from H&N35 and Global health status/QoL scale from C30. Scoring of the symptom scales/items followed the European Organisation for Research and Treatment of Cancer (EORTC) scoring manual and a linear transformation of the scores to a 0-100 point scale. Higher values are better.
Time Frame: Baseline and 5 years
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | Afatinib (BIBW 2992) | Placebo
Number analyzed (Participants) | 411 | 206
Unit on Scale
  Swallowing | 10.1 (1.00) [3.68 to NA] | 8.8 (1.12) [3.78 to NA]
  Pain HN35 | 13.1 (0.98) [1.91 to NA] | 9.9 (1.10) [3.78 to NA]
  Global health status/QoL | 29.6 (2.23) [1.87 to NA] | 33.0 (2.28) [6.21 to NA]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Placebo; Scores (swallowing scale) over time were assessed using longitudinal mixed-effects growth curve models with the average profile over time for each endpoint described by a piecewise linear model adjusted for the fixed effects baseline ECOG performance score and nodal status; Test type: Superiority or Other; p = 0.2232, Mixed Models Analysis; Degrees of freedom calculated using the Kenward-Roger method; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.81 to 3.45], Standard Error of Mean 1.08 — Afatinib minus Placebo mean adjusted for total with data for baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3)
Statistical Analysis 2: Comparison: Afatinib (BIBW 2992) vs Placebo; Scores (pain scale) over time were assessed using longitudinal mixed-effects growth curve models with the average profile over time for each endpoint described by a piecewise linear model adjusted for the fixed effects baseline ECOG performance score and nodal status; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis; Degrees of freedom calculated using the Kenward-Roger method; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [1.12 to 5.36], Standard Error of Mean 1.08 — Afatinib minus Placebo mean adjusted for total with data for baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3)
Statistical Analysis 3: Comparison: Afatinib (BIBW 2992) vs Placebo; Scores (global health/QoL) over time were assessed using longitudinal mixed-effects growth curve models with the average profile over time for each endpoint described by a piecewise linear model adjusted for the fixed effects baseline ECOG performance score and nodal status; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Degrees of freedom calculated using the Kenward-Roger method; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-5.33 to -1.49], Standard Error of Mean 0.98 — Afatinib minus Placebo mean adjusted for total with data for baseline ECOG (0 or 1) and nodal status (N0-N2a or N2b-N3)

ADVERSE EVENTS:
Time Frame: From first drug administration until 4 weeks after the last drug administration, up to 84 weeks
Arm/Group | Afatinib (BIBW 2992) | Placebo
Serious Adverse Events (participants affected / at risk) | 80/411 | 51/206
Other Adverse Events (participants affected / at risk) | 407/411 | 169/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (BIBW 2992) (N=411) | Placebo (N=206)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Retinal tear (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Disease recurrence (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Carbuncle (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 1 | 0
Hepatitis E (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 5
Respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Osteoradionecrosis (Injury, poisoning and procedural complications) | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radiation fibrosis (Injury, poisoning and procedural complications) | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Wernicke's encephalopathy (Nervous system disorders) | 1 | 0
Device occlusion (Product Issues) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (BIBW 2992) (N=411) | Placebo (N=206)
Anaemia (Blood and lymphatic system disorders) | 23 | 7
Abdominal pain (Gastrointestinal disorders) | 21 | 6
Cheilitis (Gastrointestinal disorders) | 22 | 1
Constipation (Gastrointestinal disorders) | 33 | 20
Diarrhoea (Gastrointestinal disorders) | 335 | 41
Dry mouth (Gastrointestinal disorders) | 55 | 25
Dyspepsia (Gastrointestinal disorders) | 42 | 10
Dysphagia (Gastrointestinal disorders) | 48 | 21
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 | 2
Nausea (Gastrointestinal disorders) | 43 | 24
Oral pain (Gastrointestinal disorders) | 23 | 6
Stomatitis (Gastrointestinal disorders) | 107 | 12
Vomiting (Gastrointestinal disorders) | 40 | 20
Asthenia (General disorders) | 43 | 23
Fatigue (General disorders) | 61 | 21
Mucosal inflammation (General disorders) | 126 | 17
Pyrexia (General disorders) | 29 | 7
Conjunctivitis (Infections and infestations) | 21 | 2
Nasopharyngitis (Infections and infestations) | 22 | 18
Paronychia (Infections and infestations) | 85 | 4
Upper respiratory tract infection (Infections and infestations) | 19 | 15
Weight decreased (Investigations) | 67 | 19
Decreased appetite (Metabolism and nutrition disorders) | 74 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 11
Dizziness (Nervous system disorders) | 11 | 13
Dysgeusia (Nervous system disorders) | 34 | 10
Headache (Nervous system disorders) | 18 | 12
Anxiety (Psychiatric disorders) | 10 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 30
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 22 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 54 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 | 14
Acne (Skin and subcutaneous tissue disorders) | 22 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 112 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 76 | 16
Erythema (Skin and subcutaneous tissue disorders) | 28 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 30 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 58 | 13
Rash (Skin and subcutaneous tissue disorders) | 188 | 34
Skin fissures (Skin and subcutaneous tissue disorders) | 40 | 1
Hypertension (Vascular disorders) | 18 | 12

LIMITATIONS AND CAVEATS:
The trial was stopped prematurely due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.